CLINICAL TRIAL: NCT07348770
Title: Effect of Different Cold Plasma Systems on Dental Implant Stability: A Randomized Controlled Split-Mouth Clinical Trial
Brief Title: Cold Plasma Effects on Dental Implant Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Izzet Acikan, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HRÜ/25.03.28
Record Dates: First submitted 2025-12-11; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Cold Atmospheric Plasma; Dental Implants
Keywords: Osseointegration; Surface modification; Cold atmospheric plasma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Arm (Active Comparator): The implant was inserted without the application of any supplementary surface modification.
  Interventions: Procedure: Dental implant placement
- Vacuum Plasma Application (Experimental): The implant was placed into a sterile low-pressure plasma chamber (5-10 Torr) and exposed to non-thermal low-pressure cold plasma for 60 seconds prior to placement.
  Interventions: Procedure: Dental implant placement and vacuum plasma application
- Argon Jet Plasma Application (Experimental): A portable atmospheric argon plasma jet was applied circumferentially to the implant surface for 60 seconds while the implant was rotated in a sterile holder.
  Interventions: Procedure: Dental implant placement and argon jet plasma application
- Cold Atmospheric Plasma (CAP) Application (Experimental): Cold plasma generated at atmospheric pressure using ambient air was applied circumferentially to the implant surface for 60 seconds while the implant was rotated in a sterile holder.
  Interventions: Procedure: Dental implant placement and cold atmospheric plasma application

INTERVENTIONS:
Procedure: Dental implant placement — The dental implant was placed without any plasma application.
  Arms: Control Arm
Procedure: Dental implant placement and vacuum plasma application — The dental implant was placed with non-thermal low-pressure cold plasma application
  Arms: Vacuum Plasma Application
Procedure: Dental implant placement and argon jet plasma application — The dental implant was placed with argon jet plasma application
  Arms: Argon Jet Plasma Application
Procedure: Dental implant placement and cold atmospheric plasma application — The dental implant was placed with cold atmospheric plasma application
  Arms: Cold Atmospheric Plasma (CAP) Application

SUMMARY:
Cold plasma-mediated implant surface activation may reverse the biological aging of titanium by enhancing hydrophilicity and cellular response. The aim of this study was to clinically compare the effects of three different cold plasma systems on the stability of dental implants. In this prospective randomized controlled split-mouth study, a total of 44 implants were placed in 11 patients. In each patient, four implants were randomly allocated to one of the following groups: control, vacuum plasma, argon jet plasma, and cold atmospheric plasma. All implants were placed using a single-stage protocol with a minimum insertion torque of 45 Ncm. Implant stability was assessed using resonance frequency analysis (ISQ values) immediately after placement and at 2, 4, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Presence of edentulous areas requiring ≥4 implants for fixed prosthetic rehabilitation.
* Good or moderate oral hygiene.
* Adequate patient compliance to attend all follow-up appointments.
* Willingness to voluntarily participate in the study.

Exclusion Criteria:

* Refusal to participate.
* Need for alveolar ridge augmentation.
* Systemic conditions that may impair healing (e.g., uncontrolled diabetes, immunodeficiency, ongoing chemotherapy or radiotherapy, history of head-and-neck radiotherapy, substance or alcohol abuse).
* Untreated periodontal disease.
* Heavy smoking (>10 cigarettes/day).
* Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of Implant Stability | Measurements were performed at four different time points: • Immediately after placement (baseline), • 2 weeks, • 4 weeks, • 8 weeks.
  The primary outcome measure was implant stability, quantified using Implant Stability Quotient (ISQ) values obtained by resonance frequency analysis (RFA). Changes in mean ISQ values were assessed at four predefined time points across four different implant surface treatment groups.
  The secondary outcome measure was the early stability pattern, evaluated based on serial ISQ measurements recorded during the first 8 weeks following implant placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Faculty of Dentistry, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No